CLINICAL TRIAL: NCT06976957
Title: Evaluation of the Healthcare Impact of Telemedicine Through Mobile Health App in the Follow-up and Management of Women Affected by Endometriosis (Women's eHealth And Telemedicine for Endometriosis Study - WHAT-END Study).
Brief Title: Women's eHealth And Telemedicine for Endometriosis StudyStudy).
Acronym: WHAT-END
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-TEL-2021-111
Record Dates: First submitted 2023-12-19; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis
Keywords: Endometriosis; Mobile Health; Management; Telemedicine
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Unicentric, longitudinal, prospective, experimental intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Route (No Intervention): Usual care control according to the protocol of the center for follow-up on-site visits of endometriosis affected patients.
- Telemdicine Route (Experimental): Those patients included in the intervention group will be monitored through telemedicine tools including mobile health, in addition to the usual on-site visits
  Interventions: Device: MyPlan / Movisalud App

INTERVENTIONS:
Device: MyPlan / Movisalud App — Those patients in experimental arm will be followed through a mobile app that offers different functionalities designed to improve clinical-patient communication, empower the patient in the management of his disease and treatment, detect symptoms early and individualize the interventions of professionals thanks to the patient records on the platform
  Arms: Telemdicine Route

SUMMARY:
The working hypothesis that is intended to be evaluated with this study is that the use of mobile health applications and telemedicine in the follow-up of patients affected by endometriosis offers greater satisfaction and improves the quality of care.

The patients included in the control group will be followed up according to the center's usual care protocol. Those patients included in the intervention group will be monitored through telemedicine tools including mobile health.

To evaluate the satisfaction of the application of a telemedicine program (mobile health and eConsulta) in the follow-up of the patient affected by endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic inflammatory disease that affects women where the endometrial tissue is located outside its normal location, predominantly in the pelvis, including the ovaries, pelvic ligaments and peritoneal surfaces, as well as the bladder or intestine. The presentation of the disease is diverse and ranges from superficial peritoneal lesions, ovarian endometriotic cysts, to nodules that infiltrate the tissues >5mm (deep endometriosis), all accompanied by fibrotic processes and pelvic adhesions.

The clinic of this entity is characterized by cyclical pelvic pain coinciding with menstruation, which can be accompanied by dyspareunia, dyschezia, dysuria, hematuria or rectal bleeding. In addition to the serious impact on their quality of life, these patients have much higher rates of infertility compared to the general population.

The incidence of endometriosis in the general population is difficult to quantify due to the fact that the definitive diagnosis is achieved after the direct visualization of lesions at the time of surgery, and after its anatomo-pathological study. Despite this, it is estimated that this disease affects 10% of the general population, reaching figures of 35% in symptomatic patients.

The non-specificity of the symptoms causes a diagnostic delay of approximately 8 years from the patient's first consultation, causing this disease to be detected in more advanced stages. An early diagnosis, quick access to specialized units and correct follow-up are essential to improve the quality of life of patients affected by endometriosis.

The treatments currently available for endometriosis are divided into analgesic treatments for pain control, hormonal treatments to stop the progression of the disease, and surgical treatments in patients refractory to medical treatments. Due to the fact that it is a chronic disease with the possibility of progression, the patient may require long periods of medical treatment. The side effects associated with these, the variation in response to these and the possibility of needing surgery, require a regular follow-up of these patients in the medical consultation(7,8).

Due to the need to take an anamnesis, complete physical examination and a pelvic ultrasound for the initial evaluation of the patient with suspected endometriosis, the first visit should always be done in person. Once the case has been identified and medical treatment instituted, the second visits are limited to a follow-up to assess symptoms, control adherence to treatment and the need to modify therapeutic guidelines. These follow-up visits do not require a mandatory presence and can be replaced by remote visits through information and communication technologies (ICTs).

The working hypothesis that is intended to be evaluated with this study is that the redefinition of the current care route for the patient affected by endometriosis through the incorporation of new interdisciplinary digital health tools will improve the degree of satisfaction of the users involved (patients and professionals healthcare), reduce the consumption of healthcare resources and improve the clinical management of patients.

Main objective To evaluate the satisfaction of patients affected by endometriosis after the incorporation of a follow-up program based on telemedicine (mobile health and eConsulta) by means of a randomized, longitudinal, prospective experimental, interventional clinical trial.

Secondary objectives

- To evaluate the healthcare impact of a telemedicine program (mobile health and eConsulta) in patients affected by endometriosis during follow-up in a randomized, longitudinal, prospective experimental, interventional clinical trial. Assistance impact is understood as the impact of the program on the following specific objectives:

* Reduce face-to-face care activity and consumption of health resources.
* Improve the patient's quality of life, understood as:
* Early detection of symptoms associated with clinical complications or the appearance of adverse effects associated with medication.
* Early intervention against episodes of clinical worsening.
* Reduction in the number of episodes of intense pain.
* Reduction in the intensity of pain episodes.
* Improvement of the patient's experience with regard to his pharmacological treatment (therapeutic adherence, side effects, knowledge of the therapy, discomfort of the therapy).
* Better control of lifestyles.
* Improvement of quality of life, anxiety and stress.
* Validate the sensitivity of the EQ-5D quality of life scale in endometriosis

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Patients diagnosed with endometriosis and referred for follow-up at our center and who have made at least one first face-to-face visit to the Endometriosis Unit of the HSCSP.
* That the patient has a mobile device compatible with the MyPlan web or mobile application and access to Wi-Fi or mobile data enabling the use of the technological platform from home.

Exclusion Criteria:

* Not being able to understand the nature of the study and/or the procedures to be followed.
* Not signing the informed consent.
* Be under 18 years old.
* Important language barrier.
* Lack of patient e-skills for proper use of study procedures through digital platforms.
* Impossibility of carrying out the necessary questionnaires or interviews defined in the methods of this study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the assistance received assessed through the Client Satisfaction Questionnaire (CSQ-8) | 6 months
  Patient's satisfaction with the follow-up carried out through the study period. It will be measured through the Client Satisfaction Questionnaire (CSQ-8) at the beginning and at 6 months. The Client Satisfaction Questionnaire is an 8 item measure of client satisfaction with services. The items for the CSQ-8 were selected on the basis of ratings by mental health professionals of a number of items that could be related to client satisfaction and by subsequent factor analysis. The CSQ-8 is unidimensional, yielding a homogenous estimate of general satisfaction with services. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Satisfaction with the assistance received through a 5-point Likert-type survey designed for the study | 6 months
  Patient's satisfaction with the follow-up carried out through the study period. It will be measured through a 5-point Likert-type survey designed for the study (Annex 2) at the beginning and at 6 months.

SECONDARY OUTCOMES:
Therapeutic adherence assessed through Adherence to Refills and Medications Scale (ARMS-e) questionnaire | At the beginning, at 3 and at 6 months.
  The Adherence to Refills and Medications Scale (ARMS-e) questionnaire is a validated tool designed to measure patient adherence to medication regimens, particularly focusing on refill behaviors and proper medication intake. It is widely used in clinical and research contexts to assess adherence among patients with chronic conditions or complex medication schedules. The ARMS-e is composed of items addressing difficulties patients face in obtaining and taking their medications as prescribed, including forgetfulness, understanding instructions, or logistical barriers like transportation.
  Scores for the ARMS-e range from a minimum of 12 (indicating perfect adherence with no issues) to a maximum of 48 (indicating severe non-adherence and significant challenges in following the prescribed regimen). Lower scores reflect better adherence, while higher scores suggest greater non-adherence.
Therapeutic adherence using the Haynes-Sackett questionnaire | At the beginning, at 3 and at 6 months.
  The Haynes-Sackett Questionnaire is a tool used to evaluate patient adherence to prescribed medical treatments. Commonly applied in clinical and research settings, it identifies whether patients consistently follow therapeutic recommendations. The questionnaire includes questions designed to explore patient behaviors and attitudes toward medication adherence, often addressing reasons for non-adherence and the frequency of missed doses. Scores range from 0 to 100, with 0 indicating no adherence and 100 reflecting full adherence. High scores (80-100) suggest consistent adherence, which is typically associated with better clinical outcomes. Moderate scores (50-79) indicate partial adherence, highlighting areas where improvements may be necessary. Low scores (<50) reveal significant non-adherence, which can compromise treatment effectiveness. Clinically, the Haynes-Sackett Questionnaire is used to identify barriers to adherence, such as side effects or financial challenges, design interve
Changes on quality of life (Endometriosis specific) assessed through theEndometriosis Health Profile-30 (EHP-30) | At the beginning, at 3 and at 6 months.
  The Endometriosis Health Profile-30 (EHP-30) questionnaire is a condition-specific tool designed to assess the health-related quality of life (HRQoL) in individuals with endometriosis. It captures the physical, emotional, and social impact of the condition through 30 items divided into five core domains: pain, control and powerlessness, emotional well-being, social support, and self-image. Additionally, optional modular sections address areas like work, sexual relationships, and treatment concerns, providing a comprehensive understanding of how endometriosis affects daily life.
  Each domain is scored on a scale from 0 to 100, with 0 representing the best possible HRQoL (no impact of endometriosis) and 100 indicating the worst HRQoL (severe impact). Higher scores reflect greater impairment or distress caused by endometriosis in specific areas of life.
Changes on quality of life assessed through the EuroQol5D (EQ-5D) questionnaire | At the beginning, at 3 and at 6 months.
  The EQ-5D questionnaire is a standardized instrument developed to measure health-related quality of life (HRQoL). It is widely used in clinical settings, research, and health economic evaluations to assess the impact of diseases and treatments on an individual's overall health. The EQ-5D consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has levels of severity, typically ranging from no problems to extreme problems.
  The responses are combined into a single health state that can be converted into a utility score using a scoring algorithm. Utility scores range from -0.59 to 1, where 1 indicates perfect health and 0 represents a state equivalent to death.
Number of reconsultations to the healtcare system assessed through medical assistance electronic records | at 90 and 180 days:
  Reconsultations in the healthcare system assessed through the medical assistance electronic records of the Catalan Healthcare system
Satisfaction with mobile health platform | At study completion (6 months).
  Degree of satisfaction and usability with the mobile health platform. It will be measured through an online survey designed for the different ongoing studies that are using the MyPlan platform.
Changes on Dysmenorrhoea pain scores assessed through a numerical rating scale (NRS) | At the beginning, at 3 and at 6 months.
  Level of intensity of Dysmenorrhoea (NRS 0-10), with 0 representing no pain and 10 representing the worst imaginable pain
Changes on Dyspareunia pain score assessed through a numerical rating scale (NRS) | At the beginning, at 3 and at 6 months.
  Level of intensity of Dyspareunia (NRS 0-10), with 0 representing no pain and 10 representing the worst imaginable pain
Changes on Dyschezia pain score assessed through a numerical rating scale (NRS) | At the beginning, at 3 and at 6 months.
  Level of intensity of Dyschezia (NRS 0-10), with 0 representing no pain and 10 representing the worst imaginable pain
Changes on Dysuria pain score assessed through a numerical rating scale (NRS) | At the beginning, at 3 and at 6 months.
  Level of intensity of Dysuria (NRS 0-10), with 0 representing no pain and 10 representing the worst imaginable pain
Changes on Omalgia pain score assessed through a numerical rating scale (NRS) | At the beginning, at 3 and at 6 months.
  Level of intensity of Omalgia (NRS 0-10), with 0 representing no pain and 10 representing the worst imaginable pain

CONTACTS AND LOCATIONS:
Overall Officials: Josep Estadella, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No